CLINICAL TRIAL: NCT01310049
Title: LEO 32731 - A Phase I, Single-Blind, Placebo Controlled, Single and Multiple Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Subjects
Brief Title: LEO 32731 - A Study in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: LP0058-S01
Record Dates: First submitted 2011-03-02; First posted 2011-03-07 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2011-03

CONDITIONS: Healthy Subjects
Keywords: Exploratory study in healthy subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- LP0058 oral solution (0.050 mg/mL) (Experimental): LEO 32731
  Interventions: Drug: LEO 32731
- LP0058 oral solution (0.200 mg/mL) (Experimental): LEO 32731
  Interventions: Drug: LEO 32731
- LP0058 oral solution (placebo) (Placebo Comparator): Placebo
  Interventions: Drug: LEO 32731
- LP0058 capsule 1-120 mg (Experimental): LEO 32731
  Interventions: Drug: LEO 32731
- LP0058 capsule (placebo) (Placebo Comparator): Placebo
  Interventions: Drug: LEO 32731

INTERVENTIONS:
Drug: LEO 32731 — * Part 1 and 2: Oral single dose of oral solution or capsule
  * Part 3: Twice daily dose of oral solution or capsule for 7 days

SUMMARY:
The purpose of this first-in-man trial is to determine the safety and tolerability of ascending single and multiple doses of LEO 32731 in healthy male subjects. The trial will be performed in three parts. In Part 1, single doses of LEO 32731 will be administered to healthy male subjects. In Part 2, the effect of food on the single oral dose pharmacokinetic will be investigated. In Part 3, multiple doses of LEO 32731 will be administered to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will, prior to any study related activities, have given their written informed consent to participate in the study and to abide by the study restrictions.
2. Subjects will be Caucasian males between 18 and 55 years of age and with a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive.
3. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is NOT acceptable).

Exclusion Criteria:

1. Subjects who are not, or whose partners are not willing to use appropriate contraception (such as condom) with spermicidal foam/gel/film/cream/suppository from the time of the first dose until 3 months after the final dosing occasion. Male subjects whose partners are of child-bearing potential must also agree to use an additional highly effective method of contraception
2. Subjects who have received any prescribed systemic or topical medication within 14 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
4. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
5. Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity), or a marketed drug within the past 3 months prior to the first dosing occasion.
6. Subjects who have donated any blood, plasma or platelets in 3 months prior to screening or who have made donations on more than two occasions within the 12 months preceding the first dose administration.
7. Subjects with a significant history of drug allergy as determined by the Investigator.
8. Subjects who have any clinically significant allergic disease (excluding non-active hayfever) as determined by the Investigator.
9. Subjects who have a supine blood pressure and supine pulse rate at screening higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 50 bpm, respectively
10. Subjects who consume more than 28 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits).
11. Subjects with a positive urine drug screen or alcohol breath test result at screening or first admission.
12. Subjects who smoke or who have smoked in the 3 months prior to first dose administration.
13. Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, dermatological or other major disorders as determined by the Investigator.
14. Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator.
15. Subjects who are known to have serum hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for HIV antibodies.
16. Subjects who have confirmed active/latent tuberculosis (TB).
17. Subjects who, in the opinion of their General Practitioner (GP) or the Investigator, should not participate in the study, including subjects suspected for whatever reason of not being able to comply with the requirements of the protocol.
18. Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk of participating in the study; such as QTcB interval >450 msec, 2nd or 3rd degree Atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolff-Parkinson-White Syndrome defined as PR<110 msec, confirmed by a repeat ECG.
19. Subjects who have previously taken part in or withdrawn from this study.
20. Subjects who, in the opinion of the Investigator, should not participate in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with AEs and change from baseline in vital signs (blood pressure, pulse rate and oral body temperature), ECG, telemetry and clinical laboratory. | 7 days after last dosing

SECONDARY OUTCOMES:
LEO 32731 and metabolites in blood and urine | 72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chiesa, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom